CLINICAL TRIAL: NCT02411721
Title: The Effects of Dog Intervention on Anxiety Levels in Children Undergoing an MRI Examination ; Open Label, Randomized Controlled Trail
Brief Title: The Effects of Dog Intervention on Anxiety Levels in Children Undergoing an MRI Examination
Acronym: yes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0530-14-RMB CTIL
Record Dates: First submitted 2015-03-26; First posted 2015-04-08 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Anxiety
Keywords: Anxiety; Dog Intervention; MRI; Children
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Animal assisted intervention (Experimental): The Effects of Dog Intervention on Anxiety Levels in Children. The experimental group will receive standard training on the imaging process by the MRI technician plus intervention activity with a dog
  Interventions: Behavioral: Animal Assisted Intervention
- control group (No Intervention): The control group will receive the standard training on the imaging process by the MRI technician.

INTERVENTIONS:
Behavioral: Animal Assisted Intervention — 1. Initial conversation between dog handler and child. The purpose hereof is to let the child express any fear he experiences towards the examination. The presence of the dog allows the child to project his emotions on the dog and to speak more freely about his anxiety.
  2. The dog handler informs the child on the various stages of the procedure. For this a booklet has been prepared in which a dog is the patient undergoing an MRI-scan. The child can identify with the dog in the story, and at the same time feel comforted by the dog present.
  3. Procession of emotions. The child will play freely with the dog. The purpose hereof is to create a soothing atmosphere. In stroking the soft, friendly animal the child may feel more relaxed and therefore less anxious towards the examination.
  Arms: Animal assisted intervention

SUMMARY:
Studies have shown that about two thirds of the children undergoing MRI suffer from feelings of anxiety ranging from mild apprehension to severe distress. Especially in young children, the unfamiliar surroundings, new faces, strange equipment and the noise generated during the scan, can cause feelings of stress and anxiety so severe that the test either cannot be started or cannot be performed properly due to the child's movements. For older children and adults claustrophobia is the main reason of poor image quality because of motion artifacts and/or early termination of the scan. Several studies have demonstrated the potential calming effects of companion animals on children but, to date, no formal studies on the relationship between dog intervention and children's anxiety before MRI procedures have been reported. The current study is designed to determine if dog intervention lessens children's anxiety prior to MRI

DETAILED DESCRIPTION:
MRI is an imaging method common worldwide, both for adults and children. Studies show, however, that about two thirds of the children undergoing MRI suffer from feelings of anxiety ranging from mild apprehension to severe distress. For very young children, the unfamiliar surroundings, new faces, strange equipment and particularly the noise generated during the scan, can all cause feelings of stress and anxiety so severe that the test either cannot even begin or cannot be performed properly because the child is incapable of lying still. For older children and adults claustrophobia is the main reason of poor image quality because of motion artifacts or early termination of the scan.

Anxiety is a reaction to an unfamiliar situation and its strength is far greater than the objective danger. Anxiety is characterized by subjective feelings of stress and worry that activate the autonomic nervous system.

In recent years, more and more use is made of certain techniques to prepare patients for a wide range of treatments, including methods of preparing patients for the MRI procedure, especially children. The purpose of preparation is to familiarize patients with the equipment and the stages of the imaging procedure. It also enables the technician to answer questions the patient may have and thereby avoid false assumptions about the procedure.

Intervention with animals, dogs in particular, is developing around the world and is being used in a variety of activities in rehabilitation centers, nursing homes, special education schools, hospitals and more.

In 1987 the National Institutes of Health (NIH) recognized the field of animal therapy and during the last two decades many reports have been published on the positive effects when patients interact with animals. These reports include: performance improvements, improved physiological measurements, reduction of stress and anxiety, reduced feelings of loneliness and depression, and a more speedy recovery.The animal is seen as a "friend" in the strange world of the clinic. Having a companion dog present distracts the patient from the surroundings and procedures.

In a pilot study, conducted in 2001 at the New Jersey hospital, an intervention program with a dog was introduced for reducing anxiety in adults before an MRI. This study has demonstrated that animal-assisted intervention indeed decreases the anxiety levels of patients in a pre MRI setting.

Several studies have demonstrated the potential calming effects of companion animals on children but, to date, no formal studies on the relationship between dog intervention and a child's anxiety before an MRI procedure have been reported. The current study is designed to determine if dog intervention lessens children's anxiety prior to MRI.

ELIGIBILITY:
Inclusion Criteria:

* immunocompetent children
* aged 7 to 15 years
* undergoing MRI procedures

Exclusion Criteria:

* allergy or fear of dogs
* previous Animal Assisted Invention (AAI) experience
* immunodeficiency
* asthma
* airway allergies
* open wounds
* infectious diseases that can be transferred by direct and indirect contact
* known aggressiveness

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Anxiety level | immediately after end of intervention
  To determine if among children in the experimental group the anxiety level is reduced in comparison to that of children in the control group. The State Trait Anxiety Inventory for Children (STAIC) will be used to measure the levels of anxiety of the children after the intervention / waiting period

SECONDARY OUTCOMES:
Anxiety profile assessment | up to 10 minutes after MRI scan
  To determine if, according to the assessment of the medical staff, children in the experimental group are more relaxed during the scan than children in the control group. The anxiety profile assessment will be filled out by the MRI technician who accompanies the child during the exam. The technician will be requested to rate on a scale from 1-10 the level of anxiety, the level of stress, and the state of mind of the child
Evaluate children experience | 1 week after the intervention
  To determine if one week after having undergone the scan children in the experimental group find the experience less stressful than children in the control group. A telephone questionnaire with the children will be conducted a week after the procedure in order to evaluate their experience
Quality of the MRI scan | up to two weeks after MRI scan
  To determine whether the quality of the MRI scan proves better in children in the experimental group than in children in the control group. The quality of the simulation test will be determined by the MRI physician. The criteria that will be used for determining the quality of the test are: motion artifacts and the need for repetition of the protocol due to the child's movements
Pulse measurements | Immidiately before and immediately after the intervention
  To determine if pulse rates of children in the experimental group decrease compared to those of children in the control group. Pulse measurements will be taken before and after dog intervention / waiting period.